CLINICAL TRIAL: NCT06407193
Title: Gastric Emptying Measured With MRI and Scintigraphy in Patients With Successful Versus Unsuccessful Weight Loss After Sleeve Gastrectomy
Brief Title: Gastric Emptying After Sleeve Gastrectomy
Acronym: EMRISS
Status: Recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1690
Record Dates: First submitted 2024-04-25; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gastric Emptying; Bariatric Surgery
Keywords: Gastric emptying; Gastric sleeve; MRI; Scintigraphy
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Poor weight loss group: Women aged between 20 and 55 years who underwent sleeve gastrectomy as primary procedure with TWL < 25%
  Interventions: Other: MRI and scintigraphy
- Successful weight loss group: Women aged between 20 and 55 years who underwent sleeve gastrectomy as primary procedure with TWL > 35%
  Interventions: Other: MRI and scintigraphy

INTERVENTIONS:
Other: MRI and scintigraphy — Gastric emptying measured with MRI and scintigraphy

SUMMARY:
Sleeve gastrectomy (SG) increases gastrointestinal motility, which influences feelings of fullness and satiety. By understanding the differences in gastric emptying (GE) between patients with sufficient weight loss (Total weight loss [TWL] > 35%) and insufficient weight loss (TWL < 25%), better insight in the aetiology of weight loss after sleeve gastrectomy may be obtained. GE will be measured with scintigraphy and MRI.

DETAILED DESCRIPTION:
Sleeve gastrectomy (SG) increases gastrointestinal motility, which influences feelings of fullness and satiety. Patients' weight loss response on SG varies widely and is difficult to predict. By understanding the differences in gastric emptying (GE) between patients with sufficient weight loss (Total weight loss [TWL] > 35%) and insufficient weight loss (TWL < 25%), better insight in the aetiology of weight loss after sleeve gastrectomy may be obtained. GE will be measured with scintigraphy and MRI. MRI is a non-invasive imaging method which provides more detailed images of the SG compared to the conventionally used scintigraphy scans.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 55 years who underwent sleeve gastrectomy as primary procedure with either TWL < 25% or TWL > 35%.
* Patients who had a follow-up period of 2-3 years after sleeve gastrectomy

Exclusion Criteria:

* Maximum BMI >50 kg/m2
* Patients with a disease known to affect appetite, gastric emptying or gastrointestinal motility
* Patients who are unable to stop medications that affect gastric emptying and/or motility prior to measurements. It is depending on t1/2 for how long they need to stop medication
* Patients who started menopause
* Patients with gastrointestinal problems or, gastric or intestinal diseases
* Patients with a drug or alcohol addiction
* Patients who are unable to stop smoking for 24h
* Patients who are pregnant or lactating
* Patients who have an intolerance or allergy for one of the components of the test product
* Patients who have a contra-indication to MRI scanning

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women after sleeve gastrectomy with either good or poor weight loss
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying compared between patients with poor and successful weight loss | 2-3 years
  Gastric emptying (T1/2 [min] and retention [%/min])
Gastric emptying compared between measured with MRI and scintigraphy | 2-3 years
  Gastric emptying (T1/2 [min] and retention [%/min])

SECONDARY OUTCOMES:
Sleeve characteristics compared between patients with successful and unsuccessful (poor) weight loss | 2-3 years
  Volume (sleeve size [mL] and gastric acid [mL])
to assess the association between gastric emptying rate and gastric sleeve characteristics in each group | 2-3 years
  association between outcome 1, 2 and 3
to compare subjective ratings of gastric fullness and wellbeing between patients with successful and unsuccessful weight loss | 2-3 years
  questionnaires (VAS-scale, MAIA, HADS, EBBS, Power of food scale, and Food tolerance test)

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands